CLINICAL TRIAL: NCT05335278
Title: Tolerability and Safety of Nintedanib in Myositis Associated Interstitial Lung Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Deborah Assayag, Scientist, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-5543
Record Dates: First submitted 2022-04-13; First posted 2022-04-19 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-05

CONDITIONS: Interstitial Lung Disease; Myopathy, Inflammatory
MeSH Terms: conditions — Lung Diseases, Interstitial; Myositis | interventions — nintedanib

STUDY DESIGN:
Intervention Model Description: Single group, open label study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nintedanib treatment (Experimental): Single arm treatment with nintedanib
  Interventions: Drug: Nintedanib 150 milligrams [Ofev]

INTERVENTIONS:
Drug: Nintedanib 150 milligrams [Ofev] — All patients will be given nintedanib 150 milligrams orally twice daily

SUMMARY:
There is likely a role for using anti-fibrotic medications in patients with myositis-associated interstitial lung disease (MA-ILD) to slow down disease progression, especially in patients who have fibrotic and progressive disease. These patients however are currently being excluded from clinical trials of anti-fibrotic agents in progressive ILD because of the concomitant use of immunosuppression. The benefit of anti-fibrotic agents is being assessed in other rheumatic diseases and should be assessed in MA-ILD as well. They are a unique group of patients with a heterogeneous disease, and are much more frequently on concomitant immune-modulating therapy. As such, they should be studied on their own in separate clinical trials, and the use of nintedanib should be studied as an addition to standard of care immunosuppression.

The objective of this study is to assess safety and tolerability of nintedanib in patients with MA-ILD.

ELIGIBILITY:
Inclusion Criteria:

* 1. 18 years and older 2. Diagnosis of autoimmune myopathy (dermatomyositis, polymyositis, overlap myositis or anti-synthetase syndrome) as diagnosed by a rheumatologist.

  3. Interstitial lung disease confirmed by high resolution CT scan (Extent of disease 10% or more on CT done within 12 months of enrolment) with evidence of fibrosis, defined as reticular abnormality with traction bronchiectasis with or without honeycombing.

  4. Evidence of progressive disease within 24 months of screening visit:
  1. Clinically significant decline in Forced Vital Capacity (FVC) % pred based on a relative decline of >=10%
  2. Marginal decline in FVC % pred based on a relative decline of .>=5-<10% combined with worsening of respiratory symptoms
  3. Marginal decline in FVC % pred based on a relative decline of >=5-<10% combined with increasing extent of fibrotic changes on chest imaging
  4. Worsening of respiratory symptoms such as cough or shortness of breath as well as increasing extent of fibrotic changes on chest imaging as per radiologist or pulmonologist who read the scan 5. Current and ongoing treatment with immunosuppressive medications, on a stable medication regimen and dosage for at least 6 weeks (considered standard of care medical therapy) Concomitant medications allowed are:

  <!-- -->

  1. mycophenolate,
  2. azathioprine,
  3. tacrolimus,
  4. cyclosporine,
  5. rituximab (injection within the last year),
  6. prednisone low dose =<20 mg daily,
  7. Intravenous immunoglobulins

Exclusion Criteria:

1. Contraindication to treatment with nintedanib (based on Canadian labeling)
2. The female patient is pregnant, plans to become pregnant during the course of the study, or is breastfeeding.
3. The male patient plans to father a child during the course of the study
4. Hypersensitivity to nintedanib, peanut or soy
5. Elevated liver enzymes greater than 1.5 times the upper limit of normal
6. Creatinine clearance <30 mL/min
7. Patient with risks factors of aneurysm or artery dissection, such as known history of aneurysm or uncontrolled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 11 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Tolerability - completed doses | 24 weeks
  Percentage of subjects who complete 24 weeks on nintedanib. Subjects will be considered to have completed the 24 weeks of the study if they took 90% of the study drug doses.
Safety and adverse events | 24 weeks
  numbers of patients with adverse events during course of the study

SECONDARY OUTCOMES:
Change in forced vital capacity | 24 weeks
Change in diffusion capacity of the lung for carbon monoxide | 24 weeks
Change in 6 minute walking distance | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Assayag, MD, Principal Investigator — Research Institute - McGill University Health Center
Locations (1):
- Research Institute McGill University Health Center, Montreal, Quebec, Canada